CLINICAL TRIAL: NCT05295342
Title: A Longitudinal Mixed Method Evaluation of the No Means No Intervention for Violence Prevention in Gqeberha, South Africa
Brief Title: The No Means No South Africa Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: No Means No Worldwide (Unknown)
Responsible Party: Principal Investigator, Miriam Hartmann, Principal Investigator, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0217796; REC 2/17/03/21 (Other: Human Sciences Research Council)
Record Dates: First submitted 2021-12-09; First posted 2022-03-25 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Gender-based Violence; Sexual Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Girls-only intervention arm (Experimental): Schools in this arm will receive only the girls intervention.
  Interventions: Behavioral: No Means No intervention Girls' Curriculum
- Girls and Boys intervention arm (Experimental): Schools in this arm will receive both the girls and boys intervention.
  Interventions: Behavioral: No Means No intervention Boys' Curriculum
- Control (Active Comparator): The control arm will receive the standard school-based Life Orientation curriculum.
  Interventions: Behavioral: Active comparator: Life Orientation

INTERVENTIONS:
Behavioral: No Means No intervention Girls' Curriculum — The No Means No (NMN) Girls' Curriculum is a violence prevention program designed for adolescent girls and young women 10-20 years old. This curriculum has been designed specifically for safer implementation during the COVID-19 pandemic. NMN Girls' programming is deeply rooted in Empowerment Self-Defense, which is a uniquely holistic, survivor-centered, feminist approach to self-protection skills. Youth educators called "Instructors" deliver the curriculum to young people in schools. This 8-hour intervention is comprised of classes that teach young people mental, verbal and physical self-defense skills that can be used to prevent sexual assault and other forms of gender-based violence.
  Arms: Girls-only intervention arm
Behavioral: No Means No intervention Boys' Curriculum — The No Means No (NMN) Boys' Curriculum is a violence prevention curriculum that has been designed specifically for implementation during the COVID-19 pandemic. Designed for adolescent boys and young men age 10-20. Like the girls program it is delivered by youth educators called "Instructors" in schools. This 8-hour intervention is comprised of classes that teach young people gender equitable attitudes, skills to defend equality and how to avoid violence as a power paradigm.
  Arms: Girls and Boys intervention arm
Behavioral: Active comparator: Life Orientation — The standard school-based Life Orientation curriculum
  Arms: Control

SUMMARY:
This school-based study will evaluate a behavioral intervention-the No Means No (NMN) intervention-to reduce violence among enrolled girls, ages 10-19, through a cluster-randomized control trial and a nested qualitative study.

DETAILED DESCRIPTION:
This protocol describes a mixed method evaluation study of a behavioral intervention-the No Means No (NMN) intervention-to reduce violence among enrolled girls, ages 10-19.

The No Means No intervention is an 8-12-hour behavioral intervention designed to teach Empowerment Self-Defense (ESD) to girls. A parallel intervention with boys focuses on violence perpetration by addressing issues of consent and bystander intervention. The intervention also includes a network of referrals.

The intervention will be evaluated through a cluster-randomized, controlled trial and a nested qualitative study. Implementation sites such as schools and afterschool programs (hereafter collectively referred to as schools) will be randomized to receive the girls' intervention only, the girls' and boys' interventions in parallel, or the control condition (standard of care). Control arm schools will receive the intervention as is following the study period if proven safe and effective. The study will enroll a subset of intervention participants (ages 10-19 years inclusive) at each intervention school, and an equal number of girls and boys at each control school. Experience and perpetration of sexual violence (SV), other forms of intimate partner violence (IPV), and community violence (CV) will be compared across the study arms over time, as well as engagement with referral services. At any timepoint when violence is disclosed, participants will receive first-line support and referrals for care. Participants will be followed longitudinally for 12 months.

Population: Approximately 2250 girls and 1000 boys, aged 10 to 19 years of age (inclusive) who are enrolled in 15 schools. Boys will be enrolled from the schools randomized to receive the boys' intervention and the control schools only.

Study Site(s): NMNW Implementation Site, Gqeberha, South Africa

Approach: This project will evaluate the impact of the No Means No intervention on SV prevention when paired with GBV referral services through a cluster randomized controlled study among girls and boys, with a nested qualitative component.

Study Duration: Accrual will require approximately 6 weeks. Participants in all study arms will participate in scheduled visits for enrollment (baseline), and 3, 6, and 12 months of follow-up. A subset of participants will be recruited for qualitative interviews (serial in depth interviews) to be conducted at or around 3 and 12 months post-intervention.

Primary Objectives:

1. To test the effectiveness of the No Means No intervention in reducing girls' reported experiences of sexual violence (SV);
2. To identify the mechanisms of action of No Means No on girls' reported experience of SV;

Secondary Objective:

1. To determine the effectiveness of the No Means No intervention in reducing girls' reported experiences of other forms of violence (i.e. IPV, and CV);
2. To compare the effect of simultaneous implementation of a boys violence perpetration prevention program, versus the girls' program alone or no intervention, on girls' reported experiences of SV;
3. To examine change in boys' knowledge, attitudes, and behaviors related to violence perpetration as a result of participation in a prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-19
* Enrolled in a selected school or afterschool program in the Nelson Mandela Bay municipality
* Not planning to move, de-enroll, or graduate during the study period
* Willing to participate in the 6 session No Means No intervention
* Able and willing to provide written informed consent or assent and parental consent if under 18
* English, isiXhosa, or Afrikaans speaking

Exclusion Criteria:

° Has any significant medical condition or other condition that, in the opinion of the Principal Investigator (PI)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male and female participants will enroll based on self-representation of their gender identity
Enrollment: 2173 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Change in reported sexual violence exposure incidence, intervention vs. control | Measured at baseline, six months and one year from enrollment
  Change in female participants self-report of sexual violence experience measured using adapted questions from the Manhood 2.0 study, assessed in the combined intervention arms vs. the control arm
Change in intervention mechanisms of action | Measured at three months and one year from enrollment
  Qualitative assessment of changes in theorized mechanisms of action, e.g. ways in which the intervention impacts sexual violence, explored over time using open-ended questions.

SECONDARY OUTCOMES:
Change in reported intimate partner violence exposure incidence | Measured at baseline, six months and one year from enrollment
  Change in female participants self-report of intimate partner violence experience, assessed using WHO Violence Against Women instrument (VAWI) questions in the combined intervention arms vs. the control arm
Change in reported community violence exposure incidence | Measured at baseline, six months and one year from enrollment
  Change in female participants self-report of community violence experience, assessed using questions from the Global Early Adolescent Study (GEAS) in the girls only intervention arm vs. the girls and boys intervention arm
Change in reported sexual violence exposure incidence | Measured at baseline, six months and one year from enrollment
  Change in female participants self-report of sexual violence experience measured using adapted questions from the Manhood 2.0 study, assessed in the girls-only intervention arm vs. the girls' and boys' intervention arm
Change in knowledge of sexual violence and prevention strategies | Measured at baseline, three months, six months, and one year from enrollment
  Change in self-reported knowledge of sexual violence and associated prevention strategies among male participants in the intervention vs. control arm, using questions adapted from prior evaluations (e.g. "What is consent?" and "What are the tools you can use for intervention?").
Change in gender norms | Measured at baseline, three months, six months, and one year from enrollment
  Change among male participants in gender norms according to a 20-item gender scale questions, used in the Manhood 2.0 study, in the intervention vs. control arm. Scores can range from 20 to 40 with high scores representing greater support for gender equity.
Change in attitudes towards violence | Measured at baseline, three months, six months, and one year from enrollment
  Change among male participants in attitudes towards violence according to a 4-item rape myths scale previously used in South Africa in the intervention vs. control arm. Scores can range from 4 to 12 with high scores representing lower acceptability of rape.
Change in use of intervention behaviors | Measured at baseline, three months, six months, and one year from enrollment
  Change in self-reported application of specific behaviors taught in the intervention related to violence prevention among male participants in the intervention vs. control arm, using questions from prior evaluations of the intervention, e.g. "Have you successfully intervened in any situations where someone was verbally harassing a girl or woman to stop the harassment?"
Change in sexual violence perpetration | Measured at baseline, six months and one year from enrollment
  Change in male participants who report perpetrating sexual violence in the intervention vs. control arm, measured using adapted questions from the Manhood 2.0 study.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam A Hartmann, MPH, Principal Investigator — RTI International
Locations (1):
- No Means No South Africa, Port Elizabeth, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartmann M, Mutangabende S, Nash S, Browne EN, Hatcher A, Kagesten AE, Roberts ST. Effectiveness of an empowerment-based self-defense program among South African girls: results from a cluster-randomized control trial in schools. BMC Womens Health. 2025 Mar 14;25(1):119. doi: 10.1186/s12905-025-03647-w. PMID 40087623
- See also: Website of the non-profit organization No Means No Worldwide, whose intervention is being evaluated through this trial. — https://www.nomeansnoworldwide.org/